CLINICAL TRIAL: NCT04193449
Title: Endoscopy Database for Evaluation of Predictors of Colonoscopy Outcomes
Brief Title: Colonoscopy Outcome Database
Acronym: COD
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2019/09
Record Dates: First submitted 2019-12-03; First posted 2019-12-10 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Colonoscopy Procedures
Keywords: colonoscopy; indications; outcome
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients undergoing colonoscopy: All patients' ≥18 years of age who underwent endoscopy at Portsmouth Hospitals NHS Trust, including repeat colonoscopies performed for surveillance purposes aged ≥18 in either males or females.
  Interventions: Diagnostic Test: colonoscopy

INTERVENTIONS:
Diagnostic Test: colonoscopy — colonoscopy procedure

SUMMARY:
The aim of this database is to keep routinely collected endoscopic data and outcomes in a single database which will enable the gastroenterology team to perform analyses to improve services and patient outcomes.

DETAILED DESCRIPTION:
Colonoscopy is an invasive procedure that is currently performed for a variety of reasons that centre on the detection and treatment of bowel disorders. It is time-consuming and an expensive process to develop a skilled workforce that has both the skills and the resources to provide a satisfactory colonoscopy service to the general population. Colonoscopy is also an invasive procedure associated with some serious complications like bleeding and perforation. Endoscopy resources are limited by theater space, number of endoscopes and skilled workforce. With the introduction of bowel cancer screening programmes, colonoscopy capacity has been stretched to the limit, such that extremely long waiting lists are an increasingly growing problem.

The rationale for having the database in Portsmouth is because it is a large referral centre and already has an electronic hospital endoscopy reporting system. All useful information is already stored on this platform, but the relevant clinical information is not easy to analyse in the current format. Therefore, we plan to export relevant clinical information to a database to permit retrospective data analysis. There is no need to collect any prospective data as we can achieve the desired outcomes with the current information.The research database will facilitate definitions of clinical pathways to reduce the present burden of colonoscopy on the health care system.

ELIGIBILITY:
Inclusion Criteria:

* All patients' ≥18 years of age who underwent endoscopy at Portsmouth Hospitals NHS Trust, including repeat colonoscopies performed for surveillance purposes aged ≥18 in either males or females

Exclusion Criteria:

* Patients under 18 years age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients' ≥18 years of age who underwent endoscopy at Portsmouth Hospitals NHS Trust, including repeat colonoscopies performed for surveillance purposes aged ≥18 in either males or females
Sampling Method: Non-Probability Sample
Enrollment: 23000 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Number of participants in various predicting factor's groups including sex, age, procedure indication and urgency. | 1/1/2010 to 1/1/2016.
Number of participants in different outcome groups, including normal colonoscopy, presence of pathology, and presence of interventional pathology. | 1/1/2010 to 1/1/2016.

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, Prof, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No